CLINICAL TRIAL: NCT05599308
Title: Evaluation of Blood Pressure Monitor With AFib Screening Feature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omron Healthcare Co., Ltd. (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HDV-CTD-210151
Record Dates: First submitted 2022-10-12; First posted 2022-10-31 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Prospective, parallel-cohort, open label, non-randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Atrial fibrillation (AFib) (Active Comparator): Patient with known history of AFib who are in AFib at the time of study screening.
  Interventions: Device: OMRON blood pressure monitor with AFib screening feature; Device: Microlife WatchBP Home A
- Non-Afib (Active Comparator): Patient with no known diagnosis of AFib
  Interventions: Device: OMRON blood pressure monitor with AFib screening feature; Device: Microlife WatchBP Home A

INTERVENTIONS:
Device: OMRON blood pressure monitor with AFib screening feature — Blood pressure measurement by an oscillometric blood pressure monitor
Device: Microlife WatchBP Home A — Blood pressure measurement by an oscillometric blood pressure monitor

SUMMARY:
This study aims to evaluate the safety and effectiveness of the Omron blood pressure (BP) monitor with AFib screening feature. The primary outcome is to validate if the Omron BP-monitor with AFib screening feature meets acceptance criteria in sensitivity and specificity. The acceptance criteria of the sensitivity and specificity should be statistically non-inferior to those of primary predicate device.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are eligible to participate in the study if they meet all of the following criteria. AFib participants must meet criteria 1-5. non-AFib participants must meet criteria 1-3 and 6-7.

  1. Age ≥ 22 years old
  2. Arm size within 22 cm to 42 cm in circumference
  3. Participants who have an adequate understanding about the study and have given informed written consent before participation
  4. Participants who were diagnosed with AFib and have regularly seen a cardiovascular specialist
  5. Participants who have atrial fibrillation symptoms on ECG at the time of data collection
  6. Participants who have never been diagnosed with atrial fibrillation
  7. Participants who do not have AFib symptoms on ECG at data collection time

Exclusion Criteria:

* Participants will be excluded from the study if they meet any of the following criteria.

  1. Subjects who have difficulty in ECG or blood pressure measurement due to skin rashes or wounds on the chest or arm
  2. Women who are pregnant at the time of study participation.
  3. Subjects who have had a mastectomy.
  4. Subjects with pacemakers and/or defibrillators.
  5. Subjects who have difficulty in measuring blood pressure or ECG measurements in the sitting position.
  6. Subjects who are hospitalized (in-patients)
  7. Subjects whose pulse rate is less than 40 beats/minute or more than 180 beats/minute.
  8. Subjects who have had an arterio-venous shunt or an intravascular access on either arms.
  9. Subjects who have heart failure class III or IV.
  10. Subjects who at the beginning of the scheduled study time experience any of the following newly developed conditions within the past 3 hours: chest pain, paralysis or numbness (face, arm or leg), trouble speaking or understanding, visual field loss in one or both eyes.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 574 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Sensitivity | 1 day
  To validate if the BP-monitor with AFib screening feature meets the acceptance criteria in sensitivity. Acceptance criteria is that sensitivity of the Omron BP-monitor with AFib screening feature should be statistically non-inferior to that of the primary predicate device.
Specificity | 1 day
  To validate if the BP-monitor with AFib screening feature meets the acceptance criteria in specificity. Acceptance criteria is that specificity of the Omron BP-monitor with AFib screening feature should be statistically non-inferior to that of the primary predicate device.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Accelacare of DuPage Medical Group, Winfield, Illinois
  - Accelacare of MacFarland Clinic, Ames, Iowa
  - Accelacare of Charlotte, Charlotte, North Carolina
  - Accelacare of Wilmington, Wilmington, North Carolina
  - Accelacare of Charleston, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No